CLINICAL TRIAL: NCT02767661
Title: A Phase 3 Randomized Controlled Study of Metronomic Capecitabine Combined With Aromatase Inhibitor Versus Aromatase Inhibitor Alone for First Line Treatment in Hormone Receptor-positive, Her2-negative Metastatic Breast Cancer
Brief Title: Metronomic Capecitabine Plus Aromatase Inhibitor for First Line Treatment in HR(+), Her2(-) Metastatic Breast Cancer
Acronym: MECCA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC 5010-MECCA
Record Dates: First submitted 2016-05-07; First posted 2016-05-10 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: metronomic capecitabine; aromatase inhibitor; first line treatment; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Aromatase Inhibitors; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine+Aromatase inhibitor (Experimental): Capecitabine, 500mg, orally three times daily in combination with an aromatase inhibitor (Anastrozole 1 mg, orally once daily or Letrozole 2.5mg, orally once daily or Exemestane 25mg, orally once daily)
  Interventions: Drug: Capecitabine; Drug: Aromatase Inhibitor
- Aromatase inhibitor (Active Comparator): Aromatase inhibitor (Anastrozole 1 mg, orally once daily or Letrozole 2.5mg, orally once daily or Exemestane 25mg, orally once daily)
  Interventions: Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: Capecitabine — Capecitabine, 500mg, orally three times daily (continuously)
  Other Names: xeloda
  Arms: Capecitabine+Aromatase inhibitor
Drug: Aromatase Inhibitor — Aromatase Inhibitor (Anastrozole, 1mg, orally once daily or Letrozole, 2.5mg, orally once daily or Exemestane , 25mg, orally once daily)
  Other Names: anastrozole; letrozole; exemestane

SUMMARY:
The study is designed to compare the clinical benefit following treatment with aromatase inhibitor in combination with metronomic capecitabine versus aromatase inhibitor alone in women with hormone receptor-positive, Her2-negative advanced breast cancer who have not received prior systemic anti-cancer therapies for their advanced/metastatic disease.

DETAILED DESCRIPTION:
Initial endocrine therapy (ET) is a common choice for hormone receptor positive (HR+), HER2 negative (HER2-) metastatic breast cancer (MBC) patients for its good tolerability, low toxicity and durable response. The median time to progression (TTP) of initial ET in HR+, HER2- metastatic patients is about 9 months with aromatase inhibitors (AIs). However, all metastatic patients receiving ET will develop resistance to the conventional endocrine treatments ultimately. So some novel agents, like palbociclib and everolimus, are approved to be effective in improving the efficacy of standard ET. But the fact we have to face is either palbociclib or everolimus is focusing on a single checkpoint of pathway that responsible for resistance of ET. In clinical, there are some patients without an activation of resistance-related pathways have poor response to endocrine therapy. And the mechanisms of resistance to endocrine therapy is complicated and not fully understood. So far, these novel agents have not completely solved the clinical problems of secondary drug-resistance. Maybe a broad spectrum anti-cancer therapy with low toxicity and good tolerability is more practical and promising in the near future. Metronomic chemotherapy is administration of low-dose chemotherapy to induce disease control in metastatic cancer patients, which has low-incidence of adverse effects. More and more evidences showed activity of metronomic therapy in breast cancer. Metronomic therapy with or without endocrine therapy in both metastatic and neoadjuvant setting showed considerable efficacy. Although the concept of combination of chemotherapy and endocrine therapy simultaneously was large abandoned because of previous using tamoxifen and intravenous chemotherapy showing no additional benefit, with better understanding of the biology of endocrine therapy and metronomic chemotherapy, it's worth to evaluate whether endocrine therapy plus low-dose metronomic chemotherapy brings a better clinical benefit rate without sacrificing the quality of patients' life. In this phase III study, we investigate the efficacy and safety of low-dose capecitabine plus AI to treat metastatic HR+, HER2- postmenopausal breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with locoregionally recurrent or metastatic disease not amenable to curative therapy
* Confirmed diagnosis of ER positive/Her2-negative breast cancer
* No prior systemic anti-cancer therapy for locoregionally recurrent or metastatic disease
* Any menopausal status, but premenopausal or perimenopausal patients are required to receive LHRHa treatment
* Measurable disease defined by RECIST version 1.1, or bone-only disease
* Eastern Cooperative Oncology Group (ECOG) 0-2, and life expectancy ≥ 3 months
* Adequate organ and marrow function
* Resolution of all toxic effects of prior therapy or surgical procedures

Exclusion Criteria:

* Patients who have progressed within 2 years of adjuvant endocrine therapy
* Patients who have not received prior endocrine therapy and are eligible to receive fulvestrant as initial therapy
* Patients with advanced, symptomatic, visceral spread that are at risk of life threatening complication in the short term
* Known uncontrolled or symptomatic central nervous system metastases
* Diagnosis of any other malignancy within 3 years prior to randomization (except adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ)
* Serious uncontrolled intercurrent infections or intercurrent medical or psychiatric illness

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | Baseline up to approximately 20 months
  Time from randomization to the first documentation of objective tumor progression or to death due to any cause without documented progression.

SECONDARY OUTCOMES:
Overall Survival | Baseline until death (up to approximately 48 months)
  Time from randomization to date of death due to any cause.

OTHER OUTCOMES:
Objective Response Rate (ORR) | Baseline up to approximately 20 months
  Objective response is defined as a complete response (CR) or partial response (PR) according to RECIST v.1.1. recorded from randomization until disease progression or death due to any cause.
Disease Control Rate (DCR) | Baseline up to approximately 20 months
  Disease control is defined as complete response (CR), partial response (PR), or stable disease (SD) >24 weeks according to the RECIST version 1.1 recorded in the time period between randomization and disease progression or death to any cause.
Adverse events | Baseline up to approximately 20 months
  Adverse events, serious adverse events, and laboratory tests will be analyzed and summarized according to severity.
Quality-of-life score | Baseline up to approximately 20 months
  The Functional Assessment of Cancer Therapy - Breast (FACT-B) version 4 questionnaire will be distributed to the patients by the study site personnel and will be filled out by the patients independently. Final scores (FACT-B-Total) of all subscales range from 0 to 148, where 148 represents the most favorable score and accordingly a highest QoL.
Quality-of-life score | Baseline up to approximately 20 months
  EORTC QLQ-BR23 questionnaire will be distributed to the patients by the study site personnel and will be filled out by the patients independently.

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- State Key Laboratory of Oncology in South China, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hong RX, Xu F, Xia W, Teng YE, Ouyang QC, Zheng QF, Yuan ZY, Chen DS, Jiang KK, Lin Y, Dai Z, Liu XL, Chen QJ, Wu XH, Shi YX, Huang JJ, An X, Xue C, Bi XW, Chen MT, Li H, Yao HR, Zou GR, Huang H, Zhang JM, Wang SS. Metronomic Capecitabine Plus Aromatase Inhibitor as Initial Therapy in Patients With Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Metastatic Breast Cancer: The Phase III MECCA Trial. J Clin Oncol. 2025 Apr 10;43(11):1314-1324. doi: 10.1200/JCO.24.00938. Epub 2025 Jan 2. PMID 39746176